CLINICAL TRIAL: NCT02838329
Title: The Effect of the Body Temperature 0.75% Ropivacaine on the Time to Convert Labour Epidural Analgesia to Anaesthesia for Surgical Delivery
Brief Title: Labour Epidural Top-up With Warmed Ropivacaine
Acronym: LETWR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 189493
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Epidural Top-up; Labour; Caesarian Section; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- room temperature - RT (Active Comparator): Ropivacaine used for Epidural top-up administered at room temperature
  Interventions: Drug: Ropivicaine
- body temperature BT (Experimental): Ropivacaine used for Epidural top-up administered warmed to body temperature
  Interventions: Other: warming of ropivacaine for BT; Drug: Ropivicaine

INTERVENTIONS:
Other: warming of ropivacaine for BT
  Arms: body temperature BT
Drug: Ropivicaine

SUMMARY:
The purpose of this study is to determine weather using warmed (body temperature) 0.75% Ropivicaine to convert labour epidural analgesia to surgical anaesthesia, reduces the onset time of surgical block, compared to standard room temperature

DETAILED DESCRIPTION:
In this prospective, randomised, controlled, double-blind study; parturients with functioning labour epidural analgesia requiring conversion to anaesthesia for surgical delivery (SD) - will be randomised into control and intervention groups: room temperature (RT) and body temperature (BT). The control group (RT) will receive room temperature Ropivacaine 0.75%, as is the standard practice. The treatment group (BT) will receive 0.75% Ropivicaine warmed up to 37°C temperature. Block height will be assessed every 2 minutes by a blinded investigator until the loss of sensation to cold at the level of T4, sensation to touch will be used as second modality.

Primary outcome is the time to loss of sensation to cold at T4 bilaterally as assessed with ethyl-chloride spray. Secondary outcomes will include motor block, haemodynamic stability, and use of vasopressors, shivering, sweating, nausea, pruritus, body temperature, intra-operative supplementation, and Apgar scores.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II women with an established labour epidural
* Labour analgesia with standard low-dose mixture PCEA
* Need for surgical delivery

Exclusion Criteria:

* Category 1 (crash) CS
* Spinal blockade, suggesting migration of epidural catheter
* Use of epidural bupivacaine 0.25-0.5% within 1 h
* Pyrexial parturian - ≥38°C temperature before administration of top-up
* Multiply pregnancy
* Eclampsia
* An allergy or idiosyncratic reaction to local anaesthetic
* Patient refusal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to onset of surgical anaesthesia - loss of sensation to cold at T4 bilaterally as assessed with ethyl-chloride spray. | up to 30 min

SECONDARY OUTCOMES:
Adverse effects: itching, shivering, nausea, vomiting measured on a four-point scale (0=none, 1=mild, 2=moderate, 3=severe), drop of SBP >20% of the baseline and need for vasopressors during the surgery | intraoperative
Quality of block during surgery - incidence of repeated top-up, intravenous opioids, inhaled nitrous oxide, conversion to spinal or general anaesthesia | intraoperative
Intensity of motor block - Bromage scale 3 | up to 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Kate Cheesman, MBBS, Principal Investigator — Guy's and St Thomas NHS foundation trust
Locations (1):
- St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No